CLINICAL TRIAL: NCT05954195
Title: Effect of High Intensity Interval Training in Patients With Multiple Sclerosis: Systematic Review
Brief Title: Effect of High Intensity Interval Training in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Khaled Mohamed Abdelaziz, Fatma Khaled Mohamed Abdelaziz, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HIIT in MS patients
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis AND high intensity interval training
MeSH Terms: conditions — Multiple Sclerosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: high intensity interval training starting by warm up period of 40 % from the HRmax then the interval exercise period of 85-90 % from HRmax ending by cool down period from 30 % of HRmax
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the studies mask the participants and they randomly divided into 2 groups then the care provider is masked too not to choose specific participant for specific intervention then the outcome assessor is masked to document the outcomes with fair then the investigator is masked too to document results honestly without being motivated towards the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Active Comparator): The group who received high intensity interval training
  Interventions: Other: high intensity interval training
- control/comparator group (Placebo Comparator): control group that might be placebo group, standard care group or no intervention group
  Interventions: Other: high intensity interval training

INTERVENTIONS:
Other: high intensity interval training — high intensity interval training through ergometer, with whole treatment session between 20 - 30 minutes divided into 3 parts, the 1st is warming up (40% of HRmax intensity for 2/3/5 minutes then the active training part (intervals of 85-90% of HRmax for 1 minute then rest period of 1 minute of 40 % of HRmax and so on for nearly 20 minutes ) then the last part is cooling down (30 % of HRmax for 3/5 minutes).
  Other Names: progressive aerobic training; sprinting interval exercise

SUMMARY:
In this study, we are aiming to systematically review the literature on the effect of HIIT on MS patients as improving physical performance, cognitive function, aerobic fitness and muscle strength. This could help guide the development of standardized clinical guidelines and direct clinical decision making by the physical therapists whether to implement this type of exercises or not.

DETAILED DESCRIPTION:
Multiple sclerosis patients have considerably negative effects on the community and the national and international economy. Chronic symptoms of MS such as fatigue, cognitive impairments, emotional burden and diminished physical functioning considerably affect the daily lives of people with MS and may interfere with social and quality of life factors as friendships, family relationships and occupational status. HIIT has induced significant improvements in physiological conditioning in healthy and clinical populations, and might be appropriate for persons with MS. Recently, several RCTs have been published evaluating the effect of HIIT on MS patients. Consequently, this study will systematically review all these recent literature to direct the physiotherapists whether to implement this type of exercises or not.

ELIGIBILITY:
Inclusion Criteria:

* Studies: English full texts of RCTs only, Participants: multiple sclerosis patients with age from (20-50) years old irrespectively of sex, subtype of MS, race, diagnostic criteria, community or onset of the disease, Intervention: HIIT, any comparator.

Exclusion Criteria:

* Studies other than English full text RCTs, non adults younger than 20 years and older than 50 years, populations other than multiple sclerosis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-18 (Estimated)

PRIMARY OUTCOMES:
cognitive function | 8-12 weeks or less
  serum levels of serotonin and brain derived necrotic factor (BDNF)

SECONDARY OUTCOMES:
mental processing speed | 8-12 weeks or less
  symbol digit modalities test

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abobakr Dr Alwishy, Professor, Study Chair — Physical therapy for neuromuscular disorders and its surgeries, Cairo university; Neveen Mohy-Eldin shalaby, professor, Study Chair — Faculty of medicine, Alqasr elainy, Cairo university; Hossam M. Elsaid, lecturer, Study Chair — Faculty of physical therapy of neuromuscloskeletal disorders and its surgeries, Cairo universities
Locations (1):
- Azzarqa, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
a protocol about the effect of high intensity interval training in patients with multiple sclerosis: systematic review

REFERENCES:
- [Result] Zimmer P, Bloch W, Schenk A, Oberste M, Riedel S, Kool J, Langdon D, Dalgas U, Kesselring J, Bansi J. High-intensity interval exercise improves cognitive performance and reduces matrix metalloproteinases-2 serum levels in persons with multiple sclerosis: A randomized controlled trial. Mult Scler. 2018 Oct;24(12):1635-1644. doi: 10.1177/1352458517728342. Epub 2017 Aug 21. PMID 28825348
- [Result] Langeskov-Christensen M, Grondahl Hvid L, Nygaard MKE, Ringgaard S, Jensen HB, Nielsen HH, Petersen T, Stenager E, Eskildsen SF, Dalgas U. Efficacy of High-Intensity Aerobic Exercise on Brain MRI Measures in Multiple Sclerosis. Neurology. 2021 Jan 12;96(2):e203-e213. doi: 10.1212/WNL.0000000000011241. Epub 2020 Dec 1. PMID 33262230
- [Result] Spaas J, Goulding RP, Keytsman C, Fonteyn L, van Horssen J, Jaspers RT, Eijnde BO, Wust RCI. Altered muscle oxidative phenotype impairs exercise tolerance but does not improve after exercise training in multiple sclerosis. J Cachexia Sarcopenia Muscle. 2022 Oct;13(5):2537-2550. doi: 10.1002/jcsm.13050. Epub 2022 Aug 4. PMID 35929063